CLINICAL TRIAL: NCT01678963
Title: Phase II Study of the Efficacy and Safety of Squalamine Lactate Ophthalmic Formulation 0.2% BID in Subjects With Neovascular AMD.
Brief Title: Efficacy and Safety of Squalamine Lactate Eye Drops in Subjects With Neovascular (Wet) Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohr Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OHR-002
Record Dates: First submitted 2012-08-27; First posted 2012-09-05 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: Neovascular AMD; Wet AMD; AMD; Age related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — squalamine lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Squalamine (Experimental): Squalamine eye drop 0.2%
  Interventions: Drug: Squalamine lactate
- Vehicle Control (Placebo Comparator): Eye drop vehicle control
  Interventions: Drug: Vehicle control

INTERVENTIONS:
Drug: Squalamine lactate — Ophthalmic solution 0.2%
  Arms: Squalamine
Drug: Vehicle control — Ophthalmic solution vehicle control
  Arms: Vehicle Control

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of topical ophthalmic squalamine lactate eye drops in treating patients with neovascular age-related macular degeneration (wet AMD), a degenerative retinal eye disease that causes a progressive, irreversible, severe loss of central vision.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a degenerative retinal eye disease that causes a progressive loss of central vision. AMD is the leading cause of legal blindness among adults age 50 or older in the Western world and affects 25-30 million people globally. This number is expected to triple over the next 25 years. Central vision loss from AMD is caused by the degeneration of light-sensing cells in the macula called photoreceptors. The macula, the central portion of the retina, is responsible for perceiving fine visual detail. As photoreceptors begin to degenerate, so does the individual's central vision. The extent of vision loss varies widely and is related to the type of AMD, its severity and other individual characteristics.

AMD presents itself in two different forms - a "dry" form and the more severe "wet" form. Dry AMD, the more common and milder form of AMD, accounts for 85% to 90% of all cases. It results in varying forms of sight loss and may or may not eventually develop into the wet form. Although the wet form of AMD accounts for only 10% to 15% of all AMD, the chance for severe sight loss is much greater. Wet AMD is responsible for 90% of severe vision loss associated with AMD. Approximately 500,000 new cases of wet AMD are diagnosed annually worldwide. In North America alone, approximately 200,000 new cases of wet AMD are diagnosed each year.

Squalamine lactate has been found to be an inhibitor of new blood vessel formation (angiogenesis) induced by VEGF, PDGF or bFGF. Since angiogenesis is implicated in the growth and maintenance of choroidal neovascularization, squalamine lactate is potentially an attractive development candidate in the treatment of age-related macular degeneration (AMD), in which blood vessel proliferation has a role.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age, male or female
* Have the following criteria in the study eye:

  * A diagnosis of choroidal neovascularization secondary to AMD with total lesion area ≤ 12 disc areas with CNV affecting at least 50% of the total lesion area, in at least one eye confirmed by fluorescein angiography (via the reading center)
  * Central Retinal Thickness (SD- OCT central 1 mm) of ≥ 300 um
  * Presence of sub-retinal fluid or cystoid edema on OCT. Pigment epithelial detachments without subretinal fluid or cystoid edema will be excluded
  * BCVA 20/40 to 20/230 (25 to 70 letters ETDRS)
  * If both eyes qualify the eye with the greater CRT will be the study eye. If both equal the right eye will be selected as the study eye.
* Female subjects must be 1-year postmenopausal or surgically sterilized, Women of childbearing potential must have a negative urine pregnancy test and must use an acceptable method of contraception throughout the study.
* Be willing and able to provide signed informed consent prior to participation in any study-related procedures.

Exclusion Criteria:

* Neovascularization secondary to any condition other than AMD in the study eye.
* Blood occupying greater than 50% of the AMD lesion. Blood underlying the fovea.
* Prior treatment in the study eye with bevacizumab, ranibizumab, aflibercept, PDT, submacular surgery, any antiangiogenic drug.
* Confounding ocular conditions in the study eye which will affect interpretation of OCT, VA or assessment of macular appearance eg: cataract.
* Subjects with VA worse than 20/200 (less than 34 letters) in the fellow (non-study) eye.
* Fibrosis or atrophy, retinal epithelial tear in the center of the fovea in the study eye or any condition preventing VA improvement.
* Prior ocular surgery in the study eye (Vitrectomy, scleral buckle, or glaucoma filter/shunt). Cataract surgery more than 3 months prior to enrollment is allowed so long as a posterior chamber intraocular lens is in place.
* Wearing contact lenses.
* Concomitant therapy with any drug that may affect VA, meds that may be toxic to the lens/retina or optic nerve.
* Current ocular or periocular infection in the study eye.
* Hypersensitivity to Lucentis.
* Hypersensitivity to squalamine or any component of the ophthalmic formulation
* Presence of a life threatening disease or currently on treatment for a malignancy.
* Currently on chemotherapy.
* Currently on systemic steroids.
* Pregnant or lactating.
* Investigational product use of any kind in the previous 30 days.
* Subjects for whom attendance for monthly examinations may be unreliable eg: dependent on an elderly caregiver.
* Glaucoma in the study eye (glaucomatous visual field defect and receiving treatment).
* Myocardial infarction or cerebrovascular accident or transient ischemic attacks (TIA) within the past 6 months.
* Clinical evidence of diabetic retinopathy or diabetic macular edema in the study eye.
* Uncontrolled hypertension (Diastolic BP >105 mmHg) in spite of antihypertensive medications.
* Subjects known to have HIV.
* A history of drug or alcohol abuse.
* Subjects unable to administer eye drops reliably.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Need for continued concomitant therapy | 9 months
  Lucentis (ranibizumab) is the current standard of care for the treatment of wet AMD. All patients will receive an initial injection of Lucentis prior to randomization and then be evaluated monthly for their need for further Lucentis injections using protocol defined retreatment criteria.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 9 months
  Evaluation of the effect of treatment on visual function (BCVA) as measured using the EDTRS chart measured at an initial distance of 4 meters.
Number of subjects with adverse events as a measure of safety and tolerability | 9 months
  The frequency, severity, seriousness of all adverse events including their relationship to study drug and effect on discontinuation from the study will be monitored, recorded and analysed.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Retina Associates SW, Tucson, Arizona
  - California Retinal Consultants, Bakersfield, California
  - Retina-Vitreous Associates, Beverly Hilss, California
  - Colorado Retina, Golden, Colorado
  - Florida Eye Microsurgical Institute Inc., Boynton Beach, Florida
  - Retina Health Center, Fort Myers, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Elman Retina, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vision Research Foundation, Grand Rapids, Michigan
  - Vision Research Foundation, Royal Oak, Michigan
  - Vision Research Foundation, Traverse City, Michigan
  - Total Practice Management, New Brunswick, New Jersey
  - Macula Care, New York, New York
  - Retina Associates of Cleveland, Cleveland, Ohio
  - PA Retina, Camp Hill, Pennsylvania
  - TN Retina, Nashville, Tennessee
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - University of Wisconsin, Madison, Wisconsin